CLINICAL TRIAL: NCT06462131
Title: Effectiveness of Culturally Adapted Group Cognitive Behavior Therapy on Adults With Substance Use Disorders and Their Caregivers: A Randomized Control Trial From Pakistan
Brief Title: Culturally Adapted Group Cognitive Behavior Therapy (CaGCBT-SUDs) for Substance Use Disorders and Their Caregivers
Acronym: CaGCBT-SUDs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Modern Languages (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ref No.20-16628/NRPU/R&D/HEC/
Record Dates: First submitted 2024-06-03; First posted 2024-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Treatment; Waitlist
Keywords: Group CBT; SUDs; Cultural Adaptation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- CaGCBT with TAU (Experimental): In this group, CaGCBT-SUD along with TAU will be provided.
  Interventions: Behavioral: Cultural Adapted Group cognitive Behaviroal therapy (CaGCBT)
- CBTAG with TAU and with caregivers (Active Comparator): In this group, CaGCBT-SUD along with TAU will be provided. Moreover caregivers will be provided psychoeducation
  Interventions: Behavioral: Cultural Adapted Group cognitive Behaviroal therapy (CaGCBT)
- No intervention only TAU (No Intervention): Treatment as usual

INTERVENTIONS:
Behavioral: Cultural Adapted Group cognitive Behaviroal therapy (CaGCBT) — In first session, introduction of the therapist/facilitator and group members will be made. Group rules will be discussed with members. Group members' introduction primarily focuses on participant/clients' expectations, addictive behaviors and its status, and goals. Moreover, it also emphasize on identification of any other significant issue that is contributing in burden of disease.
  Arms: CBTAG with TAU and with caregivers; CaGCBT with TAU

SUMMARY:
Pakistan is facing a massive rise in drug abuse. According to recent estimates, there are 6.7 million drug abusers, of which 4.25 million are drug dependents who need long-term treatments in residential setups. Despite these shocking statistics, there is a severe lack of evidence-based treatment, preventive measures, and drug indictment policies. Consequently, the number of drug dependents continues to increase at an alarming rate of 40,000 per year, making Pakistan one of the most drug-affected countries in the world. The ever-increasing rise in drug abuse can be devastating for a country such as Pakistan where the youth population (aged <30 years) makes up a substantial 64% of the total population. It not only affects the individual's physical and mental health but also casts devastating effects on the psycho-social and economic aspects of their lives. Adults with Substance Use Disorders (SUDs) usually come across aggravated interpersonal and family problems, loss of productivity and unemployment, poverty and crimes, overall financial problems, deaths, and accidents. Furthermore, it also destroys the norms, morality, worth, and dignity of the person's well-being and effectiveness in the growth of society. Numerous studies in Pakistan showed a lack of evidence-based treatment altogether for adults suffering from SUDs. Thus, effective interventions for SUDs that also meet the clinical reality of open treatment groups are much needed to reduce the treatment gap. Further, the implementation of evidence-based approaches like Cognitive Behavior Therapy (CBT) has an advantage with SUDs clients who are motivated. The proposed project aims at the cultural adaptation of CBT-based group intervention for adults with substance use disorders (SUDs) in Pakistan by employing a Quasi-Experimental research design, followed by Randomized Control Trials to test its effectiveness in Pakistan.

DETAILED DESCRIPTION:
Substance use has life-long impacts not only on an individual life but on their families as well. Research indicates a surge in substance use disorders in the last two decades across the globe and Pakistan has no exception. UNDP's report on drug/substance use indicates alarming prevalence rates. Furthermore, the research identifies that substance use disorder has unfavorable effects individual's quality of life and well-being. SUD places significant strain on family members and involving family caregivers in the treatment plan for opioid addiction has led to negative outcomes for the caregiver, such as depression and caregiver burden. Several researchers found that families of individuals with SUDs experience economic burden, social isolation, psychological strain, shame, embarrassment, guilt, self-blame, marital problems, and threats to their physical health. Therefore, it is important to treat SUDs as well as the burden of caregiving.

Many treatment modules have been developed to treat SUDs. Among them, group therapy was found more effective than individual therapy. CSAT lists five effective group therapy models: (1) psychoeducational groups, (2) skill development groups, (3) cognitive-behavior or problem-solving groups, (4) support groups, and (5) interpersonal groups. Furthermore, a lot of treatment modules for SUDs have been in practice. Among them, group therapy was found to be most effective in treating psychiatric or psychological issues. Furthermore, group CBT was found as effective as individual CBT. Cognitive therapy attempts to reduce excessive emotional reactions and self-defeating behaviors that are prevalent in adults with substance use disorders by modifying faulty and erroneous thinking and maladaptive beliefs that underlie these reactions. CBT for SUDs developed by Liese & Beck is based on a collaborative (trust-building), active, based on open-ended questions to a large degree, highly structured, and focused approach that gives more advantages to this therapy as compared to other therapy modalities.

Cognitive Behavior Therapy helps adults with substance use disorders to overcome their problems leading to emotional distress and helps them to visualize in a broader perspective their dependence on drugs of their choice for pleasure / or relief of discomfort. Moreover, CBT also helps to reduce the intensity and frequency of the urges by addressing their underlying beliefs and teaching them relevant techniques to not only control and manage their urges but also help them remain abstinent from the use of drugs, manage their daily life problems and thus have a more enjoyable and fulfilling life.

The following research project is based on the Cognitive-behavioral Model of problem-solving because it is a goal-directed approach that focuses on the current position of patients and mainly targets the patient's maladaptive cognitive, behavioral, and emotional patterns. Additionally, CBT techniques and planning of treatment particularly target the patient's core beliefs. If the patient's illogical beliefs change into logical and rational beliefs, the patient starts to believe that he can cope with his problems and that his problems are manageable. Core beliefs, underlying assumptions, and even the content of automatic thoughts vary across cultures. Cultural and sub-cultural backgrounds also influence beliefs about well-being, causes of illness and its cure, help-seeking behaviors, healing systems, and even the healers. The group therapy for SUDs has been developed in the West, therefore, by culturally adapting the intervention, benefits can be broadened in areas other than the West. In Pakistan, CBT has been culturally adapted for internalizing disorders such as depression and anxiety. There is a dearth of research that focuses on cultural adaptation of Group CBT especially for individuals diagnosed with SUDs.

Keeping in the backdrop to the premise, our focal point of the study would be to culturally adapt group CBT for Substance Use Disorders by Liese and Beck and to check its effectiveness on adults with substance use disorders. Further to check the effectiveness of culturally adapted CBT to treat depression and anxiety symptoms in the caregivers of SUDs in Pakistan.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed individuals with substance use disorder within the age bracket of 18-64 years.
2. In-patient of rehabilitation center and detoxified for 2 months
3. Able to give written informed consent
4. Able to read and speak Urdu

Exclusion Criteria:

1. Presence of a diagnosed physical or intellectual disability as it can prevent individuals from engaging with the intervention. This will be assessed by the research team at screening stage. Any disabilities will be identified by a relevant clinician (e.g., Psychiatrist).
2. Temporary resident unlikely to be available for follow-up
3. Being detoxified less than 2 months
4. Individuals with substance use disorder having follow up with rehabilitation center
5. Having Comorbidity with psychological disturbances like depression, anxiety etc.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Addiction Severity Index-Lite Version | Upto 8-12 weeks
  The ASI covers the following areas: medical, employment/support, drug and alcohol use, legal, family/social, and psychiatric. The ASI obtains lifetime information about problem behaviors, as well as problems within the previous 30 days. The ASI-Lite contains 22 fewer questions than the ASI, and omits items relating to severity ratings, and a family history grid. The higher a subject scores on the ASI, the greater the indication of a need for treatment.
Revised Mental Health Inventory- 5 | Upto 8-12 weeks
  The MHI-5 was developed for its use with the general population, and it includes items on psychological well-being. The total score ranges from 0 to 15, with higher scores indicating better mental health.
The Readiness to Change Questionnaire | Upto 8-12 weeks
  designed to assess stages of change in substance abusers, in terms of the Prochaska and DiClemente stages of change model. The score ranges for each scale is -10 through 0 to +10. Score towards positive end indicates patients' readiness to change.

SECONDARY OUTCOMES:
Relapse Risk Scale | Upto 8-12 weeks
  It is a 44-item self-report multidimensional instrument, which proposes to measure relapse risk among substance dependents. Lower scores indicate low risk of relapse while high scores are indicative of higher risk of relapse.
Coping Strategies Scale | Upto 8-12 weeks
  The CSS is comprised of 48 items intended to tap potential coping strategies that might be used by patients in to remain abstinent. Respondents rate the frequency (from 1 = never to 4 = frequently) of using specific strategies in the past 3 months. Total coping on the CSS was calculated by taking the mean across all 48 items.
WHO Quality of Life- Brief version | Upto 8-12 weeks
  It consists of 24 items to assess perception of quality of life in four domains, including physical health, psychological, social relationships and environment, and two items on overall QOL and general health. A higher score indicated a better quality of life.
Subjective Well-being Scale | Upto 8-12 weeks
  Subjective well-being will be measured by using following three scales: 1. PANAS (Use 5 point Likert scale to identify the positive or negative emotion experienced across week); 2. SWL(measures individuals' global cognitive judgments of their life as a whole in relation to a self-imposed ideal using five items (e.g., "In most ways my life is close to my ideal") and a seven point Likert scale (1 = strongly disagree, 7 = strongly agree); 3. HLS (assess a person's global sense of harmony in life and consists of five statements (e.g., "My lifestyle allows me to be in harmony") for which respondents are asked to indicate degree of agreement on a seven-point Likert scale (1 = strongly disagree, 7 = strongly agree).
Family Burden Interview Schedule | Upto 8-12 weeks
  It has 24 items each rated on a three-point scale: 0, no burden; 1. moderate burden; and 2, severe burden.

CONTACTS AND LOCATIONS:
Overall Officials: Anila Sadaf, PhD, Principal Investigator — NUML; Rizwana Amin, Study Director — Bahria University
Locations (5):
- Pakistan (5):
  - BMC Psychiatry, Quetta, Balochistan
  - ANF rehabilitation Centre, Islamabad, Islamabad
  - Dr. Mian Iftekhar Psychiatry Hospital, Peshawar, KPK
  - Life Care International Hospital, Lahore, Punjab Province
  - Parwarish Rehabilitation centre, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No